CLINICAL TRIAL: NCT00420030
Title: Routine Upfront Abciximab Versus Standard Peri-Procedural Therapy in Patients Undergoing Percutaneous Coronary Intervention for Cardiogenic Shock PRAGUE-7 Trial.
Brief Title: Abciximab in Patients Undergoing Percutaneous Coronary Intervention for Cardiogenic Shock
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Petr Tousek, Charles University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Charles University, Prague; MSM 0021620817
Record Dates: First submitted 2007-01-08; First posted 2007-01-09 (Estimated); Last update posted 2009-06-23 (Estimated); Status verified 2009-06

CONDITIONS: Shock, Cardiogenic
Keywords: upfront abciximab; PCI; cardiogenic shock
MeSH Terms: conditions — Shock, Cardiogenic | interventions — Abciximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Arm 1 - routine upfront administration of Reopro (Abciximab)
  Interventions: Drug: Abciximab
- 2 (Other): Reopro (Abciximab) only if needed - according to physician
  Interventions: Drug: Abciximab

INTERVENTIONS:
Drug: Abciximab — Abciximab - IIb/IIIa GP inhibitor, dosage - bolus + continuous infusion
  Other Names: Reopro

SUMMARY:
Outcome of patients with myocardial infarction complicated with cardiogenic shock is very poor. Although early mechanical revascularization has been demonstrated superior to conservative medical treatment, mortality range remains about 45-60%. Some medical registries have showed further therapeutic benefit by administration of glycoprotein (GP) IIb/IIIa inhibitors during PCI in patients with cardiogenic shock. However, there is no randomized study that supports this therapeutic strategy in these high risk patients.

Hypothesis:

GP IIb/IIIa inhibitors improve angiographic (TIMI-flow), echocardiographic (LV function) and clinical (combined end-point) outcomes in patients with myocardial infarction complicated with cardiogenic shock.

Study design:

Open "pseudorandomized" multicenter, phase IV clinical trial.

Anticipated findings:

The investigators anticipate to document better angiographic, echocardiographic and clinical outcome after upfront abciximab administration in comparison to standard periprocedural therapy in patients undergoing PCI for cardiogenic shock. This would be the first randomized clinical trial that could support this therapeutic strategy.

DETAILED DESCRIPTION:
Routine upfront abciximab versus standard peri-procedural therapy in patients undergoing percutaneous coronary intervention for cardiogenic shock PRAGUE-7 Trial.

Hypothesis:

GP IIb/IIIa inhibitors improve angiographic (TIMI-flow), echocardiographic (LV function) and clinical (combined end-point) outcomes in patients with myocardial infarction complicated with cardiogenic shock.

Study design:

Open "pseudorandomized" multicenter, phase IV clinical trial. The reason for "pseudorandomization" (i.e. randomization by even or odd date, when the PCI is performed) is ethical: it saves time, what is critical in this clinical setting. It does not delay treatment at all, while classical randomization in cardiogenic shock may sometimes delay treatment by up to 15 minutes and this is the main reason why randomized trials on shock are rarely able to enroll patients.

Groups:

Group A - Upfront administration of abciximab bolus followed by 12-hours abciximab infusion + standard therapy Group B - Standard peri-procedural therapy with possibility of abciximab administration according the interventional cardiologist. Expected rate of peri-procedural abciximab administration in this group is 20% of patients.

Allowed and excluded concomitant medication see bellow in the table

Group A Group B

Before PCI Aspirin according to physician All treatment according to Clopidogrel according to physician physician Heparin bolus 70IU/kg of body weigh Abciximab bolus 0,25 mg/kg of body weigh

During PCI Abciximab 12-hours infusion 0,125microgram/kg/min Abciximab according to Other treatment according to physician physician

Excluded Thrombolysis, Eptifibatide, Tirofiban Thrombolysis, Eptifibatide, treatment Tirofiban

Proposed sample size:

80 patients (40 patients in each group). This number of patient permit to complete the study within <2 years. Because of this and because of incidence of cardiogenic shock the study sample size is not supported statistically.

Objectives:

Primary: Thirty-day clinical combined outcome : death / reinfarction / stroke / new renal failure.

(Death = death from any cause, reinfarction = recurrent ischemic symptoms with new increase in CK-MB, stroke = any new neurologic deficit lasting > 24 hours, new renal failure = increase in creatinine to > 300 micromol/l)

Secondary: 1) Combined end-point death / reinfarction / stroke / TIMI-flow <3 / EF <30% on day 30. 2) Left ventricular EF assessed by echocardiography on the day 30 (in deceased pts. EF assumed to be 0%) 3) Rate of major bleeding complication 4) Myocardial blush score after PCI 5) TIMI-flow after PCI

Statistical analysis:

Thirty-day clinical outcome as well as other categorical characteristics of patients in the two groups will be compared by Fisher´s exact test. Group differences in continuous factors will be compared by by Student´t-test and the Wilcoxon rank-sum test.

Cardiac catheterization, PCI and abciximab:

Patients in both groups will undergo coronary angiography by femoral access using 5F or 6F sheath and catheters. All patients will receive standard antithrombotic and anticoagulant treatment either during transport or directly at the catheterization laboratory. Patients randomized into group A will receive bolus of abciximab given as a bolus dose of 0,25mg per kg of body weight immediately after randomization (either in CCU, emergency dept. or upon arrival to cath-lab), followed by an infusion of 0,125microgram/kg/min (maximum 10microgram/min) for 12 hours.

* PCI - will be performed immediately after coronary angiography if technically feasible. PCI will be performed at infarct related artery (IRA). Intracoronary stent - will be implanted if possible. Type, length and size of the stent will be choose according decision of invasive cardiologist
* Abciximab - will be given to all patients randomized into group A as mentioned above. Periprocedural abciximab bolus (0,25mg/kg) followed by 12-hours abciximab infusion (0,250 microgram/kg/min) will be given selectively to patients randomized into group B according to the decision of invasive cardiologist - we expect that GPIIb/IIIa inhibitor (abciximab) will be given to cca 10-20% of patients in this group (what is our current routine for the use of GPIIb/IIIa blockers in this setting).

Angiographic data will be stored on CD. Independent invasive cardiologist blind to clinical data and blind to the randomization of the patient, will assess TIMI flow of IRA before and after PCI (grade 0-3), myocardial blush score before and after PCI in the area of IRA (grade 0-3) and TIMI frame count after PCI.

Echocardiography:

Complete echocardiographic examination will be performed 24hours, on the day 7 and day 30 after PCI. Vivid7 ultrasound systems will be used. Data will be stored in digital form if possible (otherwise storage on S-VHS will be used). Independent observer will assess:

* end-systolic and enddiastolic diameter of left ventricle (parasternal view)
* ejection fraction measured using Simson´s method
* regional left ventricle function

Ethical consideration:

The approval of local ethical committee is required as for any other research protocol.

Anticipated finding:

We anticipate to document better angiographic, echocardiographic and clinical outcome after upfront abciximab administration in comparison to standard periprocedural therapy in patients undergoing PCI for cardiogenic shock. This would be the first randomized clinical trial that could support this therapeutic strategy.

ELIGIBILITY:
Inclusion Criteria:

1. Acute myocardial infarction (ST elevation, ST depression or bundle branch block on ECG) with indication to urgent coronary angiography
2. Signs of cardiogenic shock including incompletely developed shock (at least one of the following must be present):

   * Hypotension (BP < 90mmHg) and HR > 90/min
   * Organ hypoperfusion-cold wett sweating skin and HR>90/min
   * Need of catecholamine support to maintain BP> 90/min
   * Klip II-III + systolic BP below 120 mmHg
3. Informed consent signed either by patient or his/her relative in case of diminished consciousness.

Exclusion Criteria:

1. Contraindications for the use of abciximab, either:

   * Hypersensitiveness to Reopro components
   * Active internal bleeding
   * History of stroke in last 2 years
   * Previous history (in last 2 month) of intracranial or intraspinal surgical intervention
   * Atrio-venous malformation or aneurysm
   * Known haemorrhagic diathesis or severe uncontrolled hypertension
   * History of thrombocytopenia
   * Therapy with oral anticoagulants (warfarin)
2. Cardiogenic shock caused by severe mitral regurgitation, rupture of free left ventricle wall or interventricular septum.
3. Pre-randomization heparin dose > 10 000 U during last 6 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2006-09; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Combined end-point death/reinfarction/stroke/TIMI-flow <3/EF <30% on day 30. | 30 days

SECONDARY OUTCOMES:
Left ventricular EF assessed by echocardiography on the day 30 (in deceased pts. EF assumed to be 0%) | 30 days
Rate of major bleeding complication | 30 days
Myocardial blush score after PCI | immediately after PCI
TIMI-flow after PCI | immediatelly after PCI

CONTACTS AND LOCATIONS:
Overall Officials: Petr Widimsky, Prof,MD,PhD, Study Director — Charles University, Czech Republic; Petr Tousek, MD,PhD, Principal Investigator — Charles University, Czech Republic
Locations (1):
- Cardiocenter, University Hospital Vinohrady, Prague, Czechia

REFERENCES:
- [Derived] Tousek P, Rokyta R, Tesarova J, Pudil R, Belohlavek J, Stasek J, Rohac F, Widimsky P. Routine upfront abciximab versus standard periprocedural therapy in patients undergoing primary percutaneous coronary intervention for cardiogenic shock: The PRAGUE-7 Study. An open randomized multicentre study. Acute Card Care. 2011 Sep;13(3):116-22. doi: 10.3109/17482941.2011.567282. Epub 2011 Apr 28. PMID 21526919